CLINICAL TRIAL: NCT01455012
Title: Multicenter, Double-Blind, Placebo-Controlled, Two-Arm, Randomized, Parallel, Treatment Intervention, Sleep Lab Phase 4 Study to Assess the Effect of Rotigotine on Nocturnal Blood Pressure in Patients With Idiopathic Restless Legs Syndrome
Brief Title: Effects of Neupro on Cardiovascular Observations in Patients With Restless Legs Syndrome
Acronym: ENCORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0977; 2011-000053-23 (EudraCT Number)
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Neupro; RLS; Cardiovascular Risk; Nocturnal Blood Pressure
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine, optimal dose (minimum dose 1 mg/24 h, maximum dose 3 mg/24 h)
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — Rotigotine 1 mg/24 h, 2 mg/24 h, and 3 mg/24 h. Subjects will be titrated to their optimal/maximal dose in weekly increments of 1 mg/24 h during a Titration Period. During Maintenance Period the subjects will continue on their optimal/maximal dose for 28 days. Following the Maintenance Period, subjects will be de-escalated over 7 days, depending on their optimal/maximal dose.
  Arms: Rotigotine
Drug: Placebo — Matching Placebo. Subjects will be titrated to their optimal/maximal dose in weekly increments of 1 mg/24 h during a Titration Period. During Maintenance Period the subjects will continue on their optimal/maximal dose for 28 days. Following the Maintenance Period, subjects will be de-escalated over 7 days, depending on their optimal/maximal dose.
  Arms: Placebo

SUMMARY:
Periodic Limb Movements (PLMs) during sleep in patients with Restless Legs Syndrome (RLS) have been shown to be associated with elevations in Blood Pressure (BP). Rotigotine has been shown to effectively reduce the incidence of PLMs in patients with RLS. The current study aims to demonstrate that treatment with Rotigotine could help reduce the number of nocturnal BP elevations associated with PLMs in patients with RLS.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed and given ample time and opportunity to think about her/his participation and give her/his written informed consent
* Subject understands the investigational nature of the study and is willing and able to comply with the study requirements. Subject is willing to accept that he/she might be treated with placebo during the Treatment Period
* Subject is able to apply/remove the study patch correctly
* Subject is male or female, and is ≥18 and ≤75 years of age
* Subject meets the diagnosis of idiopathic Restless Legs Syndrome (RLS) based on the 4 essential clinical features according to the International Restless Legs Syndrome Study Group (Allen et al,2003): 1. An urge to move legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs (The urge to move can be present without uncomfortable sensations. Arms or other body parts can also be affected) 2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity, such as lying or sitting 3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues 4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present)
* Subject has a score of ≥11 on the RLS-Diagnostic Index (RLS-DI) (Benes and Kohnen, 2009)
* Subject has an initial response to previous dopaminergic treatment for RLS or has no previous dopaminergic treatment (ie, de novo)
* The subject's Body Mass Index (BMI) is ≥18 kg/m^2 and ≤35 kg/m^2
* At Baseline subject has a score of ≥15 on the IRLS (indicating moderate to severe RLS)
* At Baseline subject has a score of ≥4 points on the CGI Item 1 assessment (indicating moderately ill)
* At Baseline subject has a score of ≥15 PLM/h on the Periodic Limb Movements Index (PLMI) based on polysomnography (PSG) (recorded during the second night) as assessed by the investigator
* Subjects are on a concomitant dose of antihypertensives that is at a stable dose for at least 4 weeks prior to Baseline and hypertension is reasonably controlled while the subject agrees to continue at this dose for the duration of the study, or subject has not received concomitant treatment with antihypertensives for at least 4 weeks prior to Baseline and does not intend to start such use during the study

Exclusion Criteria:

* Subject has RLS due to renal insufficiency (uremia), iron deficiency anemia, or rheumatoid arthritis
* Subject has RLS associated with previous or concomitant therapy with dopamine D2 receptor antagonists, butyrophenones, metoclopramide, atypical antipsychotics (eg, olanzapine), tri- and tetra-cyclic antidepressants, mianserine, or lithium or H2-blockers (eg, cimetidine), or due to withdrawal from drugs such as anticonvulsants, benzodiazepines, barbiturates, and other hypnotics
* Subject has a history of sleep disturbances, such as sleep apnea syndrome (including obstructive sleep apnea), narcolepsy, sleep attacks/sudden onset of sleep, or myoclonus epilepsy either observed during PSG (local PSG evaluations) or evidenced by subject history
* Subject has uncontrolled hypertension according to the judgment of the investigator
* Subject has additional clinically relevant concomitant diseases, such as attention deficit hyperactivity disorder, polyneuropathy, akathisia, claudication, varicosis, muscle fasciculation, painful legs and moving toes, or radiculopathy
* Subject has other central nervous system diseases, such as Parkinson's disease, dementia, progressive supranuclear paresis, multisystem atrophy, Huntington's chorea, amyotrophic lateral sclerosis, or Alzheimer's disease.
* Subject has a prior history of psychotic episodes
* Subject has a history of chronic alcohol or drug abuse within the previous 12 months
* Subject has any medical or psychiatric condition, which in the opinion of the investigator, can jeopardize or would compromise the subject's ability to participate in this study
* Subject has clinically relevant cardiac dysfunction and/or arrhythmias (eg, suspected conduction system dysregulations, second or third degree atrioventricular block, complete left or right bundle branch block, sick sinus syndrome, New York Heart Association Class III or IV congestive heart failure, or had a myocardial infarction within 12 months prior to Screening [Visit 1])
* Subject has clinically relevant venous or arterial peripheral vascular disease
* Subject has a malignant neoplastic disease requiring therapy within 12 months prior to Screening (Visit 1)
* Subject is currently receiving treatment with any of the following drug classes: neuroleptics, hypnotics, antidepressants, anxiolytic drugs, anticonvulsive therapy, budipine, dopamine antagonist antiemetics (except domperidone), opioids, benzodiazepines, monoamine oxidase (MAO) inhibitors, catechol-O-methyltransferase (COMT) inhibitors, sedative antihistamines, psychostimulates, or amphetamines. If subject has received such therapy, a Washout Period of at least 7 days prior to Baseline (Visit 2) is required before starting treatment in this study
* Subject is pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined effective methods of contraception, including at least 1 barrier method, unless sexually abstinent
* Subject is a shift worker or performs other continuous non-disease-related life conditions which do not allow regular sleep at night
* At Screening Visit or Baseline Visit subject has symptomatic orthostatic hypotension
* Subject is treated with dopamine agonists within a period of 14 days prior to Baseline or L-dopa within 7 days prior to Baseline
* Subject has a medical history indicating intolerability to prior dopaminergic therapy (if pretreated)
* Subject has received previous treatment with Rotigotine
* Subject has participated in another study of an investigational drug or device within the 28 days prior to Visit 2 (Baseline) or is currently participating in another study of an investigational drug
* Subject has a known hypersensitivity to any of the components of the study medication, such as a history of significant skin hypersensitivity to adhesives, known hypersensitivity to other transdermal medications, or has unresolved contact dermatitis
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (6):
- Germany (6):
  - Berlin
  - Kassel
  - Marburg
  - München
  - Münster
  - Schwerin

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in September 2011 in order to end up with 9 German centers with enrolled subjects.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS). RS consists of all subjects randomized into this study.
Groups:
- Placebo: Placebo
  Placebo : Matching Placebo. Subjects will be titrated to their optimal/maximal dose in weekly increments of 1 mg/24 h during a Titration Period. During Maintenance Period the subjects will continue on their optimal/maximal dose for 28 days. Following the Maintenance Period, subjects will be de-escalated over 7 days, depending on their optimal/maximal dose.
- Rotigotine: Rotigotine, optimal dose (minimum dose 1 mg/24 h, maximum dose 3 mg/24 h)
  Rotigotine : Rotigotine 1 mg/24 h, 2 mg/24 h, and 3 mg/24 h. Subjects will be titrated to their optimal/maximal dose in weekly increments of 1 mg/24 h during a Titration Period. During Maintenance Period the subjects will continue on their optimal/maximal dose for 28 days. Following the Maintenance Period, subjects will be de-escalated over 7 days, depending on their optimal/maximal dose.
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 41 | 40
Completed | 30 | 36
Not Completed | 11 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Unknown reason | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS). FAS includes all randomized subjects having both a Baseline and a post-Baseline measurement for the primary efficacy variable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 29 | 37 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 6 | 11 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 56.0 (9.6) | 57.9 (10.2) | 57.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 11 | 15 | 26
Region of Enrollment [Number; unit: participants]
  Germany | 29 | 37 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Elevations of Systolic Blood Pressure (BP) During the Night That Are Associated With Periodic Limb Movements (PLMs) at the End of the 4-week Maintenance Period
Description: Polysomnography (PSG) recordings, including the assessment of continuous Blood Pressure and 12-lead Electrocardiogram (ECG), were obtained on 2 consecutive nights prior to Baseline Visit and prior to End of Maintenance Period (Visit 7) for up to 8 hours per night. Readings from the first night of the PSG were only used for analysis if the PSG from the second night was determined to be not valid for evaluation. Influence of Periodic Limb Movements (PLMs) on sleep is reflected in the Periodic Limb Movement-Related Arousal Index (PLMAI). Arousal is defined as sudden change in the EEG activity and the index illustrates to what degree the PLMs contribute to arousal from sleep. Sleep stages and time spent in each sleep stage were determined from Electroencephalogram (EEG) readings.
  A negative value in Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: Full Analysis Set (FAS) includes all randomized subjects having both a Baseline and a post-Baseline measurement for the primary efficacy variable. All 66 subjects in the FAS are included in the analysis of this Outcome Measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Nocturnal Elevations of Systolic BP
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
Nocturnal Elevations of Systolic BP | -79.61 (189.3) [-119.25 to -39.97] | -239.95 (237.1) [-275.34 to -204.56]
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; The 95 % Confidence Interval (CI) and the p-value for the mean difference between Rotigotine and Placebo was obtained from a linear Analysis of Covariance (ANCOVA) model with fixed effects for treatment and Baseline antihypertensive use and a covariate for the Baseline number of nocturnal elevations of Systolic Blood Pressure that are associated with Periodic Limb Movements (PLMs); Test type: Superiority or Other; p < 0.0001, ANCOVA — The analysis of this primary efficacy variable was performed using a two-sided alpha level of 5 %; Mean Difference (Final Values) = -160.34, 95% CI 2-sided [-213.23 to -107.45], Standard Error of Mean 26.46 — The treatment effect was estimated on the basis of the Least Square Mean (LSM) of the difference as well as on the 95 % Confidence Interval and the p-value for that difference. Difference to Placebo was calculated as Rotigotine-Placebo

2. Secondary Outcome: Change From Baseline in the Total Number of Elevations of Systolic Blood Pressure (BP) During the Night at the End of the 4-week Maintenance Period
Description: as for outcome 1
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nocturnal Elevations of Systolic BP
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
Nocturnal Elevations of Systolic BP | -34.3 (243.4) | -199.8 (262.8)

3. Secondary Outcome: Change From Baseline in the Periodic Limb Movements Index (PLMI) at the End of the 4-week Maintenance Period
Description: The PLMI is defined as Periodic Limb Movements (PLMs)/ total time in bed in hours. PLMs are measured by Polysomnography (PSG). A negative value in PLMI Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Periodic Limb Movements/hour
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
Periodic Limb Movements/hour | -15.2 (50.3) | -50.1 (44.5)

4. Secondary Outcome: Change From Baseline in the International Restless Legs Syndrome Rating Scale (IRLS) at the End of the 4-week Maintenance Period
Description: The IRLS is a subject-based scale that consists of 10 items to evaluate the severity of major RLS symptoms and the impact of the disease on subjects' daytime functioning. Each of the 10 items is measured on a scale that ranges from 0 (not present) to 4 (severe). A sum score between 0 (no RLS symptoms present at all) and 40 (maximum severity in all symptoms) across all 10 items was calculated. A negative value in IRLS Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -12.5 (9.0) | -18.5 (8.0)

5. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-Quality of Life (RLS-QoL) at the End of the 4-week Maintenance Period
Description: The RLS-QoL is a disease-specific instrument for the evaluation of Quality of life. It consists of 12 items and the overall sum score is calculated from all 12 items and measured on a scale that ranges from 0 (lowest Quality of life) to 60 (highest level of Quality of life). A negative value in RLS-QoL Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -11.0 (11.9) | -17.8 (13.2)

6. Secondary Outcome: Clinical Global Impressions (CGI) Item 2 (Change of Condition) at the End of the 4-week Maintenance Period
Description: The CGI Item 2 score measures any change in severity of RLS from Baseline on a 7-point scale consisting of the following categories:
  * 1- Very much improved
  * 2- Much improved
  * 3- Minimally improved
  * 4- No change
  * 5- Minimally worse
  * 6- Much worse
  * 7- Very much worse
Time Frame: At the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
participants
  Very much improved | 9 | 26
  Much improved | 9 | 7
  Minimally improved | 4 | 3
  No change | 6 | 1
  Minimally worse | 1 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0

7. Secondary Outcome: Clinical Global Impressions (CGI) Item 1 (Severity of Illness) at the End of the 4-week Maintenance Period
Description: The CGI Item 1 score measures the severity of illness on a 7-point scale consisting of the following categories:
  * 1- Normal, not ill at all
  * 2- Borderline ill
  * 3- Mildly ill
  * 4- Moderately ill
  * 5- Markedly ill
  * 6- Severely ill
  * 7- Among the most extremely ill subjects
Time Frame: At the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
participants
  Normal, not ill at all | 2 | 6
  Borderline ill | 8 | 18
  Mildly ill | 7 | 9
  Moderately ill | 8 | 2
  Markedly ill | 3 | 2
  Severely ill | 1 | 0
  Among the most extremely ill subjects | 0 | 0

8. Secondary Outcome: Clinical Global Impressions (CGI) Item 3 (Therapeutic Efficacy) at the End of the 4-week Maintenance Period
Description: The CGI Item 3 score measures the therapeutic efficacy on a 4-point scale consisting of the following categories:
  * 1- Very good
  * 2- Moderate
  * 3- Slight
  * 4- Unchanged or worse
Time Frame: At the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
participants
  Very good | 11 | 31
  Moderate | 10 | 4
  Slight | 3 | 1
  Unchanged or worse | 5 | 1

9. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 1 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 1 measures subject's satisfaction with sleep on a 11-point scale that ranges between 0 (completely satisfied) to 10 (completely dissatisfied). The ratings are given by the subjects. A negative value in RLS-6 Item 6 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -3.4 (3.1) | -4.1 (3.3)

10. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 2 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 2 measures the severity of RLS at time falling asleep on a 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects. A negative value in RLS-6 Item 2 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -3.9 (3.3) | -4.6 (3.8)

11. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 3 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 3 measures the severity of RLS during the night on a 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects. A negative value in RLS-6 Item 3 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -3.7 (3.5) | -4.9 (3.3)

12. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 4 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 4 measures the severity of RLS during day rest on a 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects. A negative value in RLS-6 Item 4 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -2.7 (3.4) | -2.9 (2.9)

13. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 5 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 5 measures the severity of RLS during day not rest on a 11-point scale that ranges between 0 (none) to 10 (very severe). The ratings are given by the subjects. A negative value in RLS-6 Item 5 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -1.3 (1.9) | -1.3 (2.6)

14. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 Rating Scales (RLS-6) Item 6 at the End of the 4-week Maintenance Period
Description: The RLS-6 consists of 6 items of which four items are designed to assess severity of RLS and two items cover sleep and daytime tiredness. Item 6 measures subject's tiredness or sleepiness during the day on a 11-point scale that ranges between 0 (not at all) to 10 (very severe). The ratings are given by the subjects. A negative value in RLS-6 Item 6 Change from Baseline indicates an improvement from Baseline. The higher the negative value the better the improvement.
Time Frame: Baseline to the end of the 4-week Maintenance Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 37
units on a scale | -2.5 (2.8) | -3.5 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 16 weeks from Screening Period to the Safety Follow-Up Visit.
Description: Adverse Events refer to the Safety Set consisting of all randomized subjects who received at least one dose of study medication.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 19/40 | 23/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rotigotine (N=40)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 6 (6) | 5 (5)
Application site pruritus (General disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (5) | 7 (8)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 7 (8)
Somnolence (Nervous system disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days